CLINICAL TRIAL: NCT03642912
Title: Coagulation Monitoring in Patients on Extracorporeal Membrane Oxygenation Hämostaseologisches Monitoring Bei Patienten Mit Extrakorporaler Membranoxygenierung
Brief Title: Coagulation Monitoring in Patients on Extracorporeal Membrane Oxygenation (Observational Study)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Michael Zoller MD, Principal Investigator, Ludwig-Maximilians - University of Munich
Other Study IDs: LMU 18-047
Record Dates: First submitted 2018-08-11; First posted 2018-08-22 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Coagulation and Hemorrhagic Disorders; Extracorporeal Membrane Oxygenation Complication
Keywords: ECMO; haemostasis; coagulation; haemostatic alterations
MeSH Terms: conditions — Thrombosis; Hemorrhagic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ECMO patients: ECMO patients treated on the intensive care units of the Department of Anesthesiology of LMU Munich

SUMMARY:
Coagulation disorders are on top of the list of extracorporeal-membrane oxygenation (ECMO) complications. They contribute significantly to morbidity and mortality of ECMO patients. This observational study aims to evaluate coagulation profiles of ECMO patients treated on the intensive care units of the Department of Anaesthesiology of LMU Munich.

DETAILED DESCRIPTION:
Coagulation disorders are on top of the list of extracorporeal-membrane oxygenation (ECMO) complications. They contribute significantly to morbidity and mortality of ECMO patients. This observational study aims to evaluate coagulation profiles of ECMO patients treated on the intensive care units of the Department of Anaesthesiology of LMU Munich. Adult ECMO patients are included in the study after informed consent.

Bleeding and thromboembolic complications as well as treatment details are recorded. Additional coagulation laboratory markers (such as von-Willebrand-factor, ADAMTS13-protease, platelet function tests and thromboelastometric tests) are correlated with clinical signs of bleeding. Regular ultrasound examination of the large vessels are performed to Screen for thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* patient treated on ICU of Department of Anesthesiology of LMU Munich
* treated with ECMO
* age >/= 18 years (adult patients only)
* informed consent

Exclusion Criteria:

* underage patients
* pregnant patients
* hemoglobin level < 8mg/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: critically ill patients treated with ECMO
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
platelet function parameter | after starting ECMO therapy - up to 28 days after starting ECMO therapy
  platelet function test
platelet function parameter | one week after ending ECMO therapy
  platelet function test
coagulation parameter | after starting ECMO therapy - up to 28 days after starting ECMO therapy
  thromboelastometric test
coagulation parameter | one week after ending ECMO therapy
  thromboelastometric test

SECONDARY OUTCOMES:
inflammatory parameter | after starting ECMO therapy - up to 28 days after starting ECMO therapy
  bradykinin levels
inflammatory parameter | one week after ending ECMO therapy
  bradykinin levels

OTHER OUTCOMES:
bleeding assessment | after starting ECMO therapy - up to 28 days after starting ECMO therapy
  all patients are screened for signs of bleeding or thrombosis
bleeding assessment | one week after ending ECMO therapy
  all patients are screened for signs of bleeding or thrombosis

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zoller, MD, Principal Investigator — Department of Anaesthesiology, LMU Munich; Mathias Bruegel, MD, Principal Investigator — Institute of Laboratory Medicine, LMU Munich; Dominik J Hoechter, MD, Study Director — Department of Anaesthesiology, LMU Munich; Michael Weigand, MD, Study Director — Institute of Laboratory Medicine, LMU Munich; Bernhard Zwißler, MD, Prof., Study Chair — Department of Anaesthesiology, LMU Munich; Daniel Teupser, MD, Prof., Study Chair — Institute of Laboratory Medicine, LMU Munich
Locations (1):
- Department of Anesthesiology, LMU Munich, Munich, Germany

IPD SHARING:
Plan to Share IPD: No
sharing individual participant data is restricted by EU General Data Protection Regulation (GDPR)